CLINICAL TRIAL: NCT04840680
Title: Post-Marketing Surveillance (Usage Results Study) of Ixazomib Citrate in Patients With Multiple Myeloma in South Korea
Brief Title: A Study of Real-World Use of Ixazomib Citrate in People With Multiple Myeloma (MM)
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: C16030
Record Dates: First submitted 2021-04-09; First posted 2021-04-12 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Multiple Myeloma
Keywords: Drug Therapy
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants With MM: Participants with MM who are newly prescribed and will start treatment with ixazomib citrate in a real-world clinical practice setting will be observed prospectively for up to 6 years 11 months.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study.

SUMMARY:
In this study, people with MM will be treated with ixazomib citrate according to their clinic's standard practice. The main aim of the study is to check for side effects from ixazomib citrate.

DETAILED DESCRIPTION:
This is a non-interventional, prospective, observational post-marketing surveillance study of ixazomib citrate in participants with MM.

The study will assess the safety and effectiveness of ixazomib citrate for its approved indications in a clinical practice setting under real-world conditions.

The study will enroll approximately 165 participants. The data will be prospectively collected, at the centers from medical files and recorded into electronic case report forms (e-CRFs).

All participants will be enrolled in a single observational group:

• Participants With MM

The study will be conducted in South Korea. The overall duration of the study will be approximately 6 years and 11 months. Data will be collected over and up to a 6 months-surveillance period (per participant) once enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with MM.
2. Participants who are prescribed and initiate ixazomib citrate for the treatment of MM according to the ixazomib citrate South Korean product label.

Exclusion Criteria:

1. Participants treated with ixazomib citrate outside of the locally approved label in South Korea.
2. Participants for which ixazomib citrate is contraindicated as per product label.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with MM who have been newly prescribed with ixazomib citrate in routine clinical practical setting will be observed prospectively.
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Up to 6 months

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | From first administration of study drug to the date of disease progression or death due to any cause, whichever occurs first (up to 6 months)
  PFS is defined as the estimated length of time since the start of treatment with ixazomib to disease progression (PD), study end or death, whichever occurs first. PFS will be assessed by International Myeloma Working Group (IMWG) Criteria, PD: increase of greater than or equal to (>=) 25 percent (%) from lowest response value in any one or more of the following: serum M-component increase >=0.5 gram per deciliter (g/dL) or urine M-component increase >=200 milligram (mg)/24-hour; difference between involved and uninvolved free light chains (FLC) levels increase must be greater than (>) 10 mg/dL; bone marrow plasma cell >=10%; definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas; development of hypercalcemia that can be attributed solely to plasma cell proliferative disorder. PFS will be analyzed using Kaplan-Meier method.
Overall Response Rate (ORR) | Up to 6 months
  ORR is defined as the percentage of participants with stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR) based on the review of the myeloma response data assessed by IMWG criteria. sCR: CR as defined below plus normal FLC ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence; CR: negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and less than (<) 5% plasma cells in bone marrow; VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or >=90% reduction in serum M-protein plus urine M-protein level <100 mg/24 hour; PR: >=50% reduction of serum M-protein and >=90% reduction in urine M-protein or <200 mg/24 hour, or >=50% decrease in uninvolved FLC or >=50% reduction in plasma cells. At baseline, a >=50% decrease in size of soft tissue plasmacytomas is required.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (20):
- South Korea (20):
  - Hallym University Sacred Heart Hospital, Anyang
  - SOONCHUNHYANG UNIVERSITY HOSPITAL Bucheon, Bucheon-si
  - Inje University Busan Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Keimyung University Dongsan Hospital, Daegu
  - Chungnam National Unversity Hospital, Daejeon
  - Chonnam National University Hwasun Hospital, Hwasun
  - The Catholic University of Korea, Incheon ST. Marys Hospital, Incheon
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Samsung medical center, Seoul
  - The Catholic University of Korea Seoul ST. Mary's Hospital, Seoul
  - Chung-Ang University Hospital, Seoul
  - Ewha womans university medical center, Seoul
  - Korea University Guro Hospital, Seoul
  - Ajou University Hospital, Suwon
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju
  - Yongin Severance Hospital, Yŏngin

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/60768b60688ad8001f42fb94